CLINICAL TRIAL: NCT03489031
Title: Basal Study - Observational Multicentric Clinical Study: Basal Insulin And Compensation Glycemic In Diabetic Patients In Basal Bolus Outpatient.
Brief Title: Basal Insulin And Compensation Glycemic In Diabetic Patients In Basal Bolus Outpatient.
Acronym: BASAL
Status: Completed | Type: Observational
Sponsor: Associazione Medici Endocrinologi (Other)
Responsible Party: Sponsor
Other Study IDs: BASAL Study
Record Dates: First submitted 2018-03-20; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetes Mellitus, Type 1: patients with type 1 diabetes
- Diabetes Mellitus, Type 2: patients with type 2 diabetes

SUMMARY:
Multicentric, observational, cross-sectional study in Italy. The aims are to evaluate the basal/total ratio of daily insulin dose (b/T) in diabetic outpatients type 1 (T1) and type 2 (T2) on basal-bolus regimen, by investigating whether there is a relationship with HbA1c and episodes of hypoglycemia.

DETAILED DESCRIPTION:
The study was commissioned by the Italian Association of Clinical Endocrinologists (Associazione Medici Endocrinologi - AME) and approved by the Ethical Committee of Cuneo Hospital (BASAL Study- OSS 001/2016 - rif ENDO 30). The research was open to all specialists taking care of patients with diabetes in Italy.

The primary endpoint was glycemic control, evaluated by HbA1c levels, according to b/T.

Secondary endpoints were occurrence of major hypoglycemic episodes according to b/T; differences between patients with T1 and T2.

An ad hoc form was developed and used to record all medical findings. The form was emailed to all participating centers who then emailed or faxed it back to our data manager. Data were checked for accuracy.

The following data were required: age, gender, body weight and height, country of origin, type of diabetes and its duration, units of basal and total (basal plus prandial) daily insulin, type of basal insulin (Glargine, Detemir or Degludec), use and dosage of metformin, and number of major hypoglycemic episodes (<40 mg/dL or requiring caregivers intervention) in the last three months. Serum creatinine and HbA1c levels obtained within the previous two months were also required.

Each participating center recruited between 20 and 40 diabetic outpatients. Inclusion criteria were as follows: adult outpatients (≥20 and ≤80 years) with T1 or T2 diabetes mellitus, on basal-bolus insulin regimen (basal insulin, i.e. Glargine, Detemir or Degludec, plus at least two prandial insulin shots) for at least six months, usually assuming three daily meals, and capable of informed consent.

ELIGIBILITY:
Inclusion Criteria:

* adult outpatients (≥20 and ≤80 years);
* T1 or T2 diabetes mellitus;
* basal-bolus insulin regimen (basal insulin, i.e. Glargine, Detemir or Degludec, plus at least two prandial insulin shots) for at least six months;
* assuming three daily meals;
* capable of informed consent.

Exclusion Criteria:

* pregnancy;
* breast-feeding;
* severe liver or renal failure (eGFR <30 mL/min/1.73 m2);
* use of OADs (except for metformin);
* hospitalization for any cause in the last six month;
* glucocorticoid treatment in the last six month;
* oncologic treatment in the last six month;
* Ramadan in the last six months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All diabetic patients respecting eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 1036 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
basal/total ratio | last six month
  To evaluate the basal/total ratio of daily insulin dose (b/T) in diabetic outpatients type 1 (T1) and type 2 (T2) on basal-bolus regimen

SECONDARY OUTCOMES:
glycaemic control | last six month
  relationship between b/T ratio and HbA1c
hypoglycemia | last six month
  relationship between b/T ratio and episodes of hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Borretta, MD, Principal Investigator — Associazione Medici Endocrinologi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heinemann L, Heise T, Wahl LC, Trautmann ME, Ampudia J, Starke AA, Berger M. Prandial glycaemia after a carbohydrate-rich meal in type I diabetic patients: using the rapid acting insulin analogue [Lys(B28), Pro(B29)] human insulin. Diabet Med. 1996 Jul;13(7):625-9. doi: 10.1002/(SICI)1096-9136(199607)13:73.0.CO;2-2. PMID 8840095
- [Result] Laubner K, Molz K, Kerner W, Karges W, Lang W, Dapp A, Schutt M, Best F, Seufert J, Holl RW. Daily insulin doses and injection frequencies of neutral protamine hagedorn (NPH) insulin, insulin detemir and insulin glargine in type 1 and type 2 diabetes: a multicenter analysis of 51 964 patients from the German/Austrian DPV-wiss database. Diabetes Metab Res Rev. 2014 Jul;30(5):395-404. doi: 10.1002/dmrr.2500. PMID 24302583
- [Result] Nosek L, Roggen K, Heinemann L, Gottschalk C, Kaiser M, Arnolds S, Heise T. Insulin aspart has a shorter duration of action than human insulin over a wide dose-range. Diabetes Obes Metab. 2013 Jan;15(1):77-83. doi: 10.1111/j.1463-1326.2012.01677.x. Epub 2012 Sep 9. PMID 22882249
- [Derived] Castellano E, Attanasio R, Giagulli VA, Boriano A, Terzolo M, Papini E, Guastamacchia E, Monti S, Aglialoro A, Agrimi D, Ansaldi E, Babini AC, Blatto A, Brancato D, Casile C, Cassibba S, Crescenti C, De Feo ML, Del Prete A, Disoteo O, Ermetici F, Fiore V, Fusco A, Gioia D, Grassi A, Gullo D, Lo Pomo F, Miceli A, Nizzoli M, Pellegrino M, Pirali B, Santini C, Settembrini S, Tortato E, Triggiani V, Vacirca A, Borretta G; all on behalf of Associazione Medici Endocrinologi (AME). The basal to total insulin ratio in outpatients with diabetes on basal-bolus regimen. J Diabetes Metab Disord. 2018 Oct 1;17(2):393-399. doi: 10.1007/s40200-018-0358-2. eCollection 2018 Dec. PMID 30918874